CLINICAL TRIAL: NCT05341739
Title: A Phase II Study of Pre-Operative Stereotactic Radiosurgery Followed by Surgical Resection for Brain Metastases
Brief Title: A Phase II Study of Pre-Op SRS Followed by Surgical Resection for Brain Metastases
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Allegheny Singer Research Institute (also known as Allegheny Health Network Research Institute) (Other)
Collaborators: Elekta Limited (Industry)
Responsible Party: Principal Investigator, Rodney Wegner, Radiation Oncologist, Allegheny Singer Research Institute (also known as Allegheny Health Network Research Institute)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-240-AGH
Record Dates: First submitted 2022-04-18; First posted 2022-04-22 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-03

CONDITIONS: Brain Metastases, Adult
Keywords: Stereotactic Radiosurgery (SRS)
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Pre-Operative Stereotactic Radiosurgery (SRS) (Experimental): Subjects are treated using the standard of care SRS to a total dose of 24-27 Gray (Gy) in 3 fractions with a once daily fractionation or every other day at treating physician discretion. The preferred dose will be 27 Gy, with ability to drop dose down to 24 Gy if normal tissue constraints cannot be met. It should be noted, that while the dosing remains within standard of care, the timing of the radiation (pre-operative) is still not considered standard of care but is supported by emerging data as described in the study background. Additional metastatic lesions may be treated using SRS according to institutional practices. The radiation dose prescribed to the non-index lesions is at the discretion of the treating physicians. Surgical resection will be performed within 2 weeks of completion of SRS.
  Interventions: Other: Pre-operative Stereotactic Radiosurgery

INTERVENTIONS:
Other: Pre-operative Stereotactic Radiosurgery — Pre-operative SRS will be performed prior to the surgical resection of the brain metastases.

SUMMARY:
This is a research study to determine if performing stereotactic radiosurgery (SRS) prior to surgical resection of the brain metastasis (tumor) will improve local control, in other words, increase the possibility of total removal of the primary tumor without local recurrence on longterm follow up. This research study will also determine if pre-operative SRS will lower the risk of radionecrosis that is the breakdown of body tissue at the original tumor site, and the development of leptomeningeal disease.

DETAILED DESCRIPTION:
Patients with a solid tumor malignancy that has metastasized to the brain are invited to participate in this trial. Upon enrollment to this study a subject will undergo stereotactic radiosurgery (SRS) using the Elekta Gamma Knife Icon, being treated in once daily 15 minute fractions of 9 Gray (Gy) or every other day 15 minute fractions of 9 Gy for a total dose of 27 Gy in 3 doses. A subject will undergo a routine CT and MRI simulation to determine positioning of the head prior to the start of the SRS treatment. Within two (2) weeks after completion of SRS a subject will undergo a routine surgical resection of the brain metastasis. Prior to the SRS treatment and during the follow up phase of the study MRIs will be performed, which are standard of care. Subjects will also complete a quality of life questionnaire. The duration of subject's time participating in this study is 2 years.

ELIGIBILITY:
Inclusion Criteria:

1. Histologic proof or unequivocal cytologic proof of solid tumor malignancy. This may be obtained from either the primary site or any metastatic site
2. Solid tumor brain metastases
3. Age≥ 18 years
4. Karnofsky Performance Status ≥70
5. Patient must have agreed to undergo surgical resection to manage at least 1 brain metastasis
6. Maximum tumor diameter of index lesions <5 cm. (Index lesion defined as the brain metastasis which will undergo surgical resection)
7. Brain MRI within 1 month of initiation of brain SRS
8. No prior whole brain radiotherapy (WBRT) or radiation therapy directed to index brain metastases
9. Patients of childbearing potential (male or female) must practice adequate contraception due to possible harmful effects of radiation therapy on an unborn child
10. Patient must have the ability to understand and the willingness to sign a written informed consent document
11. All patients must be informed of the investigational nature of this study and must be given written informed consent in accordance with institutional and federal guidelines
12. Patients receiving prior SRS for brain metastases in other locations of the brain are eligible
13. Patients with multiple brain metastases planned for surgical intervention are eligible for this study. Each individual brain metastasis will be treated

Exclusion Criteria:

1. Prior WBRT or SRS to the index lesion
2. Brain metastasis greater than or equal to (≤) 5 cm in maximum diameter
3. Patients must not have a serious medical or psychiatric illness that would in the opinion of the treating physician prevent informed consent or completion of protocol treatment, and/or follow-up visits.
4. Karnofsky Performance Status (KPS) less than (<)70.
5. Patients with absolute contraindication to MRI imaging are not eligible for the study
6. Patients who are pregnant are excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-12-14 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Radiographic Local Control | 4-5 Years from first subject enrolled.
  Radiographic local control at 1 year following completion of pre-operative SRS followed by surgical resection of brain metastasis. Local control will be according to the Response Assessment criteria for Neuro-Oncology (RANO) for brain metastases.

SECONDARY OUTCOMES:
Leptomeningeal disease | 4-5 years from first subject enrolled.
  MRI will be utilized to evaluate for evidence of leptomeningeal spread at 3 month intervals following preoperative SRS followed by surgical resection of the brain metastasis.
Radio-Necrosis | 4-5 years from first subject enrolled
  Pathologic confirmation of radio-necrosis will be recorded as binary variable for each patients as well as the date of surgery confirming radio-necrosis, as applicable.
Pseudo-Progression | 4-5 years from first subject enrolled
  Defined as worsening T1 post-gadolinium contrast enhancement and fluid attenuated inversion recovery (FLAIR) changes following SRS which resolve independently without any intervention beyond steroids.

CONTACTS AND LOCATIONS:
Overall Officials: Rodney E Wegner, MD, Principal Investigator — AHN Radiation Oncology
Locations (1):
- Allegheny General Hospital, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No